CLINICAL TRIAL: NCT02702973
Title: Characteristic Analysis of Retinopathy Associated With High Doses of Interferon α-2b Therapy in Patients With Melanomas of the Skin
Brief Title: Characteristic Analysis of Retinopathy Associated With High Doses of Interferon α-2b Therapy
Acronym: CARI2b
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: 2016WD2M1
Record Dates: First submitted 2016-02-18; First posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-02

CONDITIONS: Retinopathy
Keywords: Characteristic analysis
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Observational Model: Case-Crossover
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observe the fundus characteristics: Observe the fundus characteristics after high doses of interferonα-2b therapy in patients with melanomas of the skin.
  Interventions: Other: Observe the fundus characteristics after therapy.

INTERVENTIONS:
Other: Observe the fundus characteristics after therapy.

SUMMARY:
The high doses of interferon α-2b therapy in patients with melanomas of the skin may induced retinopathy, especially in the patients with hypertension or diabetes, so these patients should be followed up after treatment.

DETAILED DESCRIPTION:
Patients with melanomas of the skin whose tumors have been resected completely were collected. The detailed ocular examinations including intraocular pressure, slit lamp microscope, indirect ophthalmoscope and color fundus photography were done before the induction therapy, 2 weeks after the induction therapy, after the whole course of induction therapy and each month in the maintenance treatment period. Fundus examinations were carried out by experienced ocular fundus doctors and the retinopathy characteristics were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, at least 18 years of age.
2. ECOG performance status 0 or 1.
3. Patients must have histologically confirmed stage IB to stage III primary melanoma of cutaneous origin (AJCC 7th edition classification).
4. Must complete all primary therapy (wide excision with or without lymphadenectomy).

Exclusion Criteria:

1. Mucous membrane or ocular melanoma.
2. Any evidence of distant metastasis (CT-scan of brain, Chest X ray or CT, abdominal ultrasound or CT and ultrasound of regional lymph nodes at screening).
3. Patients with retinopathy on baseline fundoscopic examination at the start of interferon therapy.
4. History of any other malignancy within the last ten years (except basal cell carcinoma or squamous cell carcinoma of the skin and carcinoma in situ of the cervix).
5. Patients with severe cardiac disease (e.g. NYHA Functional Class III or IV, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina), severe liver disease or severe renal disease.
6. Patients who have a history of depression or other psychiatric diseases requiring hospitalisation.
7. History or presence of autoimmune disease (i.e. autoimmune hepatitis, thyroid auto-immune dysfunction, systemic lupus erythematodes),
8. Unwilling or unable to comply with the requirements of the protocol for the duration of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eighteen patients with melanomas of the skin whose tumors have been resected completely were collected
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Change of ocular fundus after high doses of interferon α-2b therapy at the 1st week. | the 1st week

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin University,No.1 Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Lan S, Cui Z, Yin Q, Liu Z, Liang L, He H, Liu H, Guo Z, Yu Y, Wu D. Prospective study of clinical characteristics of melanoma patients with retinopathy caused by a high-dose interferon alpha-2b. Melanoma Res. 2021 Dec 1;31(6):550-554. doi: 10.1097/CMR.0000000000000769. PMID 34524220